CLINICAL TRIAL: NCT02640404
Title: Safety of a Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) in Healthy Subjects Aged 9 Months to 55 Years in Vietnam
Brief Title: Safety of a Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine in Healthy Subjects in Vietnam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA90; U1111-1143-9207 (Other: WHO)
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; Menactra®; Meningococcal Vaccine
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Menactra® Vaccine (9 to 23 Months) (Experimental): Participants (infants and toddlers) received 2-dose series of study vaccine with 3-month interval (first dose at Day 0 and second dose 3 months after dose 1).
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine
- Menactra® Vaccine (2 to 55 Years) (Experimental): Participants (children, adolescents and adults) received 1 dose of study vaccine at Day 0.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular. 2 doses 3 months apart
  Other Names: Menactra®
  Arms: Menactra® Vaccine (9 to 23 Months)
Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular.
  Other Names: Menactra®
  Arms: Menactra® Vaccine (2 to 55 Years)

SUMMARY:
The aim of the study is to assess the safety of Menactra vaccine in infants, toddlers, children, adolescents, and adults

Objective:

* To describe the safety profile after each and any dose (when applicable) of Menactra vaccine in participants aged 9 months to 55 years for registration.

DETAILED DESCRIPTION:
Infants and toddlers will receive 2 doses of vaccine 3 months apart. Children ≥ 2 years through adults aged 55 years will receive 1 dose of vaccine. All participants will be evaluated for safety up to 28 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 months to 55 years on the day of the first study visit
* For adults: Informed consent form had been signed and dated by the participant For minors: Informed consent form had been signed and dated by the parent or legally acceptable representative. In addition, in accordance with the Independent Ethics Committee /Institutional Review Board requirements and as appropriate for the age of the participant, the participant may be required to sign and date the informed consent form if aged 12 to 17 years or assent form if aged 8 to 11 years
* Participant and/or parent/legally acceptable representative (if applicable) were able to attend all scheduled visits and to comply with all study procedures

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following study vaccination
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (>=2 mg/kg/day prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substances
* Laboratory-confirmed, self-reported, or known (as reported by the parent/legally acceptable representative) thrombocytopenia, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Personal history of Guillain-Barré syndrome
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 37.5°C or ≤ 35.5°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event had subsided
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction

Ages: 9 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 224 (Actual)
Dates: Start 2016-06-06; Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Asia Pacific
Locations (1):
- Vĩnh Long, Vinh Long Province, Vietnam

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 06 June 2016 through 16 June 2016 at a single center in Vietnam.
Pre-assignment Details: A total of 224 participants (112 for each group) were enrolled and vaccinated in the study.
Groups:
- Menactra® Vaccine (9 to 23 Months): Participants (infants and toddlers) received 2 doses of 0.5 mL Menactra® Vaccine, intramuscularly, with 3-month interval (first dose at Day 0 and second dose, 3 months after dose 1).
- Menactra® Vaccine (2 to 55 Years): Participants (children, adolescents and adults) received 1 dose of 0.5 mL Menactra® Vaccine, intramuscularly at Day 0.
Period: Overall Study
Arm/Group | Menactra® Vaccine (9 to 23 Months) | Menactra® Vaccine (2 to 55 Years)
Started | 112 | 112
Completed | 110 | 112
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Vaccine (9 to 23 Months) | Menactra® Vaccine (2 to 55 Years) | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Customized [Count of Participants; unit: Participants]
  9 to 23 months | 112 | 0 | 112
  2 to 11 years | 0 | 43 | 43
  12 to 17 years | 0 | 33 | 33
  18 to 55 years | 0 | 36 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 57 | 109
  Male | 60 | 55 | 115
Region of Enrollment [Number; unit: participants]
  Vietnam | 112 | 112 | 224

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection-Site Reactions Following Vaccination: Menactra® Vaccine (9 to 23 Months)
Description: Solicited injection (Inj.) site reactions: Tenderness/Pain (Grade 1: minor reaction when Inj. site touched; Grade 2: cries/protests when Inj. site touched; Grade 3: cries when injected limb moved, or the movement of the injected limb is reduced), Erythema and Swelling (Grade 1: >0 to <25 mm, Grade 2: >=25 to <50 mm, Grade 3: >=50 mm). Number of participants with any of the Grade 1, 2 or 3 solicited injection-site reactions and Grade 3 solicited injection-site reactions were reported.
Time Frame: Within 7 days post-vaccination 1, Within 7 days post-vaccination 2
Population: Safety analysis set included all participants who received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Menactra® Vaccine (9 to 23 Months)
Number analyzed (Participants) | 112
Participants
  Any Inj. site pain (post-vaccination 1) | 15
  Grade 3 Inj site pain (post-vaccination 1) | 0
  Any Inj site pain (post-vaccination 2): number analyzed (Participants) | 110
  Any Inj site pain (post-vaccination 2) | 15
  Grade 3 Inj site pain (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Inj site pain (post-vaccination 2) | 0
  Any Erythema (post-vaccination 1) | 1
  Grade 3 Erythema (post-vaccination 1) | 0
  Any Erythema (post-vaccination 2): number analyzed (Participants) | 110
  Any Erythema (post-vaccination 2) | 2
  Grade 3 Erythema (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Erythema (post-vaccination 2) | 0
  Any Swelling (post-vaccination 1) | 1
  Grade 3 Swelling (post-vaccination 1) | 0
  Any Swelling (post-vaccination 2): number analyzed (Participants) | 110
  Any Swelling (post-vaccination 2) | 2
  Grade 3 Swelling (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Swelling (post-vaccination 2) | 0

2. Primary Outcome: Number of Participants Reporting Solicited Injection-Site Reactions Following Vaccination: Menactra® Vaccine (2 to 55 Years)
Description: Solicited injection (Inj.) site reactions in children (2-11 years), adolescents and adults (12-55 years): Tenderness/Pain (Grade 1: easily tolerated [children], no interference with activity [adolescents and adults]; Grade 2: sufficiently discomforting [children], some interference[adolescents and adults]; Grade 3: unable to perform usual activities[children]; significant interference with daily activities [adolescents and adults]), Erythema and Swelling (Grade 1: >0 to<25 mm [children], >=25 to <=50 mm [adolescents and adults]; Grade 2: >=25 to <50 mm [children], >=51 to <=100 mm [adolescents and adults], Grade 3: >=50 mm [children]; >100 mm[adolescents and adults]). Number of participants with any of Grade 1, 2 or 3 solicited injection-site reactions and Grade 3 solicited injection-site reactions were reported.
Time Frame: Within 7 days post-vaccination
Population: Safety analysis set included all participants who received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Menactra® Vaccine (2 to 55 Years)
Number analyzed (Participants) | 112
Participants
  Any Inj site pain | 28
  Grade 3 Inj site pain | 1
  Any Erythema | 2
  Grade 3 Erythema | 0
  Any Swelling | 1
  Grade 3 Swelling | 0

3. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactions Following Vaccination: Menactra® Vaccine (9 to 23 Months)
Description: Solicited systemic reactions: Fever (Grade 1: >=38.0 degree Celsius to <=38.5 degree Celsius; Grade 2: >38.5 degree Celsius to <=39.5 degree Celsius; Grade 3: >39.5 degree Celsius), Vomiting (Grade 1: 1 episode per 24 hours, Grade 2: 2-5 episodes per 24 hours, Grade 3: >=6 episodes per 24 hours), Crying abnormal (Grade 1: <1 hour; Grade 2: 1-3 hours; Grade 3: >3 hours), Drowsiness (Grade 1: sleepier than usual or less interested in surroundings; Grade 2: Not interested in surroundings or did not wake up for a feed / meal; Grade 3: Sleeping most of the time or difficult to wake up), Appetite loss (Grade 1: eating less than normal; Grade 2: missed 1 or 2 feeds / meals completely; Grade 3: refuses >=3 feeds / meals or refuses most feeds / meals), Irritability (Grade 1: easily consolable; Grade 2: requiring increased attention; Grade 3: inconsolable). Number of participants with any of the Grade 1, 2 or 3 systemic reactions and Grade 3 systemic reactions were reported.
Time Frame: Within 7 days post-vaccination 1, Within 7 days post-vaccination 2
Population: Safety analysis set included all participants who received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Menactra® Vaccine (9 to 23 Months)
Number analyzed (Participants) | 112
Participants
  Any Fever (post-vaccination 1) | 9
  Grade 3 Fever (post-vaccination 1) | 1
  Any Fever (post-vaccination 2): number analyzed (Participants) | 110
  Any Fever (post-vaccination 2) | 9
  Grade 3 Fever (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Fever (post-vaccination 2) | 0
  Any Vomiting (post-vaccination 1) | 8
  Grade 3 Vomiting (post-vaccination 1) | 0
  Any Vomiting (post-vaccination 2): number analyzed (Participants) | 110
  Any Vomiting (post-vaccination 2) | 10
  Grade 3 Vomiting (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Vomiting (post-vaccination 2) | 1
  Any Crying Abnormal (post-vaccination 1) | 9
  Grade 3 Crying Abnormal (post-vaccination 1) | 0
  Any Crying Abnormal (post-vaccination 2): number analyzed (Participants) | 110
  Any Crying Abnormal (post-vaccination 2) | 8
  Grade 3 Crying Abnormal (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Crying Abnormal (post-vaccination 2) | 1
  Any Drowsiness (post-vaccination 1) | 6
  Grade 3 Drowsiness (post-vaccination 1) | 0
  Any Drowsiness (post-vaccination 2): number analyzed (Participants) | 110
  Any Drowsiness (post-vaccination 2) | 5
  Grade 3 Drowsiness (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Drowsiness (post-vaccination 2) | 0
  Any Appetite lost (post-vaccination 1) | 22
  Grade 3 Appetite lost (post-vaccination 1) | 0
  Any Appetite lost (post-vaccination 2): number analyzed (Participants) | 110
  Any Appetite lost (post-vaccination 2) | 17
  Grade 3 Appetite lost (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Appetite lost (post-vaccination 2) | 0
  Any Irritability (post-vaccination 1) | 13
  Grade 3 Irritability (post-vaccination 1) | 1
  Any Irritability (post-vaccination 2): number analyzed (Participants) | 110
  Any Irritability (post-vaccination 2) | 7
  Grade 3 Irritability (post-vaccination 2): number analyzed (Participants) | 110
  Grade 3 Irritability (post-vaccination 2) | 1

4. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactions Following Vaccination: Menactra® Vaccine (2 to 55 Years)
Description: Solicited systemic reactions: Fever (Grade 1: >=38.0 degree Celsius to <=38.4 degree Celsius; Grade 2: >=38.5 degree Celsius to <=38.9 degree Celsius; Grade 3: >=39.0 degree Celsius), headache, malaise and myalgia (Grade 1: no interference with activity, Grade 2: some interference, Grade 3: significant interference). Number of participants with any of the Grade 1, 2 or 3 systemic reactions and Grade 3 systemic reactions were reported.
Time Frame: Within 7 days post-vaccination
Population: Safety analysis set included all participants who received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Menactra® Vaccine (2 to 55 Years)
Number analyzed (Participants) | 112
Participants
  Any Fever | 5
  Grade 3 Fever | 1
  Any Headache | 17
  Grade 3 Headache | 3
  Any Malaise | 24
  Grade 3 Malaise | 1
  Any Myalgia | 20
  Grade 3 Myalgia | 1

ADVERSE EVENTS:
Time Frame: Non-serious Adverse Events (AEs) data were collected from Day 0 up to 28 days post-vaccination. Serious adverse event data were collected from Day 0 throughout the study (up to 135 days for participants 9 to 23 months of age and up to 28 days for participants 2 to 55 years of age).
Description: A solicited reaction is an AE that is prelisted in the electronic case report form (eCRF) and considered to be related to vaccination. A solicited reaction is therefore an adverse drug reaction (ADR) observed and reported under the conditions (nature and time to onset) prelisted (i.e., solicited) in the eCRF. An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or time to onset post-vaccination.
Arm/Group | Menactra® Vaccine (9 to 23 Months) | Menactra® Vaccine (2 to 55 Years)
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/112
Serious Adverse Events (participants affected / at risk) | 16/112 | 0/112
Other Adverse Events (participants affected / at risk) | 86/112 | 49/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menactra® Vaccine (9 to 23 Months) (N=112) | Menactra® Vaccine (2 to 55 Years) (N=112)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 3 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 2 | 0
Febrile convulsion (Nervous system disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Menactra® Vaccine (9 to 23 Months) (N=112) | Menactra® Vaccine (2 to 55 Years) (N=112)
Gastrointestinal disorder (Gastrointestinal disorders) | 13 | 0
Vomiting (Gastrointestinal disorders) | 18 | 1
Crying (General disorders) | 15 | 0
Injection site pain (General disorders) | 23 | 28
Malaise (General disorders) | 0 | 24
Pyrexia (General disorders) | 24 | 7
Bronchiolitis (Infections and infestations) | 11 | 0
Bronchitis (Infections and infestations) | 8 | 1
Nasopharyngitis (Infections and infestations) | 24 | 0
Pharyngitis (Infections and infestations) | 6 | 4
Respiratory tract infection (Infections and infestations) | 12 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 3
Decreased appetite (Metabolism and nutrition disorders) | 32 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 20
Headache (Nervous system disorders) | 0 | 17
Somnolence (Nervous system disorders) | 8 | 0
Irritability (Psychiatric disorders) | 16 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.